CLINICAL TRIAL: NCT00003991
Title: Multi-Center, Randomized Open-Label Study to Evaluate the Safety and Efficacy of Immunotherapy With Subcutaneous Maxamine (Histamine Dihydrochloride) Plus Proleukin (Interleukin-2) Versus No Treatment (Standard of Care) in Patients With Acute Myeloid Leukemia in First or Subsequent Complete Remission (CR)
Brief Title: Interleukin-2 Plus Histamine Dihydrochloride in Treating Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Maxim Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000067196; MAXIM-MP-MA-0201; CWRU-MAXI-1998
Record Dates: First submitted 1999-11-01; First posted 2004-06-03 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2011-12

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia in remission
MeSH Terms: conditions — Leukemia | interventions — aldesleukin; Histamine

INTERVENTIONS:
Biological: aldesleukin
Drug: histamine dihydrochloride

SUMMARY:
RATIONALE: Interleukin-2 may stimulate a person's white blood cells to kill acute myeloid leukemia cells. Histamine dihydrochloride may prolong remission and reduce the risk of relapse in patients with acute myeloid leukemia in remission.

PURPOSE: Randomized phase III trial to determine the effectiveness of interleukin-2 plus histamine dihydrochloride in treating patients who have acute myeloid leukemia that is in remission following previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the efficacy of interleukin-2 plus histamine dihydrochloride (Maxamine) vs no further therapy in prolonging the leukemia free survival in patients with acute myeloid leukemia in first or subsequent complete remission (CR) following consolidation therapy. II. Compare the relapse rate, overall survival, and quality of life in this patient population treated with interleukin-2 plus Maxamine vs no further therapy. III. Compare the remission inversion rate in patients in subsequent CR with this treatment regimen vs no further therapy.

OUTLINE: This is a randomized, open label, parallel, multicenter study. Patients are stratified according to complete remission (first vs subsequent). Patients are randomized to one of two treatment arms. Arm I: Following consolidation chemotherapy or autologous stem cell transplantation, patients receive interleukin-2 subcutaneously followed by histamine dihydrochloride subcutaneously over 5-7 minutes twice daily on days 1-21. Treatment repeats every 6 weeks for 3 courses and then every 9 weeks for 7 courses in the absence of disease relapse or unacceptable toxicity. Arm II: Patients receive no further therapy following consolidation chemotherapy or autologous stem cell transplantation. Quality of life is assessed prior to study, and at visits 6, 7, 10, 11, 16, 17, and 22. Patients are followed for relapse and survival every 3 months for 2.5 years.

PROJECTED ACCRUAL: A total of 360 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Cytologically confirmed acute myeloid leukemia (AML) in first complete remission (CR) or subsequent CR Less than 5% blasts in normal bone marrow Less than 3 months since last dose of chemotherapy OR Less than 6 months since achieving CR

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: WHO 0-1 OR Karnofsky 70-100% Life expectancy: Greater than 3 months Hematopoietic: WBC at least 1,500/mm3 Platelet count at least 75,000/mm3 Hepatic: PTT normal Bilirubin no greater than 2 times upper limit of normal (ULN) SGOT and SGPT no greater than 2 times ULN Renal: Creatinine no greater than 1.5 times ULN Cardiovascular: No class III or IV heart disease No hypotension, severe hypertension, or serious or uncontrolled cardiac dysrhythmia (e.g., ventricular arrhythmias) No acute myocardial infarction within the past 12 months No active uncontrolled angina pectoris No symptomatic arteriosclerotic blood vessel disease Pulmonary: No history of asthma within the past 5 years Other: No other active malignancies except localized basal or squamous cell skin cancer or carcinoma in situ of the cervix HIV negative No prior or active peptic or esophageal ulcer disease No history of hypersensitivity to histamine or histamine products, or severe allergies Not pregnant or nursing

PRIOR CONCURRENT THERAPY: Biologic therapy: Prior autologous stem cell transplantation allowed No prior allogeneic stem cell transplantation No other concurrent immunomodulating agents Chemotherapy: See Disease Characteristics Prior induction or consolidation therapy allowed No concurrent chemotherapy Endocrine therapy: At least 24 hours since prior corticosteroids No concurrent steroids Radiotherapy: Not specified Surgery: Not specified Other: No concurrent alternative therapy (e.g., laetrile, Brudzinski's treatment, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 1998-07; Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Berryhill, Study Chair — Maxim Pharmaceuticals
Locations (118):
- United States (32):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - Arizona Cancer Center, Tucson, Arizona
  - Scripps Clinic, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Kaiser Permanente-Southern California Permanente Medical Group, San Diego, California
  - Sidney Kimmel Cancer Center, San Diego, California
  - Pacific Hematology/Oncology, San Francisco, California
  - Bethesda Bone Marrow Stem Cell Transplant Institute, Boynton Beach, Florida
  - University of Florida Health Science Center - Jacksonville, Jacksonville, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas
  - Oncology and Hematology Associates, Westwood, Kansas
  - Maine Center for Cancer Medicine and Blood Disorders, Scarborough, Maine
  - Henry Ford Hospital, Detroit, Michigan
  - Providence Hospital Cancer Center, Southfield, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Nevada Cancer Center, Las Vegas, Nevada
  - Nevada Medical Group-Internal Medicine, Reno, Nevada
  - University of New Mexico Cancer Research & Treatment Center, Albuquerque, New Mexico
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - Our Lady of Mercy Medical Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Ireland Cancer Center, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - West Clinic, P.C., Memphis, Tennessee
  - Boston Cancer Group, Memphis, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Cancer Care Institute of South Texas, San Antonio, Texas
  - South Texas Cancer Institute, San Antonio, Texas
- Australia (16):
  - Liverpool Hospital, Liverpool, New South Wales
  - Newcastle Mater Misericordiae Hospital, Newcastle, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - St. Vincent's Hospital, Sydney, New South Wales
  - NSW Breast Cancer Institute, Westmead, New South Wales
  - Wesley Clinic for Hematology/Oncology, Auchenflower, Queensland
  - Royal Brisbane Hospital, Brisbane, Queensland
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Mater Public Hospital, South Brisbane, Queensland
  - Hanson Center for Cancer Research, Adelaide, South Australia
  - Queen Elizabeth Hospital, Adelaide, South Australia
  - Monash Medical Center, East Bentleigh, Victoria
  - Peter MacCallum Cancer Institute, East Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Royal Perth Hospital, Perth, Western Australia
  - Fremantle Hospital, Fremantle
- Canada (8):
  - Vancouver General Hospital, Vancouver, British Columbia
  - Queen Elizabeth II Health Science Center, Halifax, Nova Scotia
  - London Health Sciences Centre, London, Ontario
  - Ottawa Regional Cancer Center - General Division, Ottawa, Ontario
  - Seaforth Medical Centre, Montreal, Quebec
  - Hopital Du Sacre-Coeur de Montreal, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Pavillion de Quebec, Québec, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
- Denmark (2):
  - Aalborg Hospital, Aalborg
  - Odense University Hospital, Odense
- Estonia (2):
  - Tallinn Central Hospital, Tallinn
  - University of Tartu, Tartu
- Finland (4):
  - Helsinki University Central Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
  - Tampere University Hospital, Tampere
  - Turku University Central Hospital, Turku
- France (8):
  - Centre Hospitalier Regional et Universitaire d'Angers, Angers
  - CHR de Besancon - Hopital Jean Minjoz, Besançon
  - Hopital Beaujon, Clichy
  - Hopital Andre Mignot, Le Chesnay
  - Centre Hospitalier Regional de Lille, Lille
  - Hopital Edouard Herriot, Lyon
  - CHR Hotel Dieu, Nantes
  - Centre Henri Becquerel, Rouen
- Germany (16):
  - Zentralklinikum Augsburg, Augsburg
  - Universitaetsklinikum Charite, Berlin
  - Evang. Diakonissenanstalt, Bremen
  - Medizinische Klinik I, Dresden
  - Universitaetsklinik und Strahlenklinik - Essen, Essen
  - Klinikum der J.W. Goethe Universitaet, Frankfurt
  - Martin Luther Universitaet, Halle
  - Universitats-Krankenhaus Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Medizinische Klinik und Poliklinik, Heidelberg
  - Staedtische Kliniken Osnabruek, Osnabrück
  - Universitat Rostock, Rostock
  - Caritasklinik St. Theresa, Saarbrücken
  - Universitaetsklinikum Tuebingen, Tübingen
  - Klinikum der Universitaet Ulm, Ulm
  - Medizinische Poliklinik der Universitat, Würzburg
- Israel (6):
  - Rambam Medical Center, Haifa
  - Hadassah University Hospital, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Kaplan Hospital, Rehovot
  - Tel-Aviv Medical Center-Ichilov Hospital, Tel Aviv
- New Zealand (5):
  - University of Auckland School of Medicine, Auckland
  - Canterbury Health Laboratories, Christchurch
  - Waikato Hospital, Hamilton
  - Palmerston North Hospital, Palmerston North
  - Wellington Hospital, Wellington
- Sweden (16):
  - County Hospital (Malar Hospital), Eskilstuna
  - Sahlgrenska University Hospital, Gothenburg (Goteborg)
  - County Hospital/Kalmar, Kalmar
  - Central Hospital, Karlstad
  - University Hospital of Linkoping, Linköping
  - Lund University Hospital, Lund
  - Malmo University Hospital, Malmo
  - Regional Hospital, Örebro
  - County Hospital (Karnsjukhuset), Skövde
  - Huddinge Hospital, Stockholm
  - Karolinska Hospital, Stockholm
  - County Hospital/Sundsvall, Sundsvall
  - County Hospital/Uddevalla, Uddevalla
  - Umea Universitet, Umeå
  - University Hospital - Uppsala, Uppsala
  - County Hospital/Vasteras, Västerås
- United Kingdom (3):
  - Birmingham Heartlands and Solihull NHS Trust (Teaching), Birmingham, England
  - Leeds Teaching Hospital Trust, Leeds, England
  - Manchester Royal Infirmary, Manchester, England

REFERENCES:
- [Result] Buyse M, Michiels S, Squifflet P, Lucchesi KJ, Hellstrand K, Brune ML, Castaigne S, Rowe JM. Leukemia-free survival as a surrogate end point for overall survival in the evaluation of maintenance therapy for patients with acute myeloid leukemia in complete remission. Haematologica. 2011 Aug;96(8):1106-12. doi: 10.3324/haematol.2010.039131. Epub 2011 May 5. PMID 21546500
- [Result] Buyse M, Squifflet P, Lucchesi KJ, Brune ML, Castaigne S, Rowe JM. Assessment of the consistency and robustness of results from a multicenter trial of remission maintenance therapy for acute myeloid leukemia. Trials. 2011 Mar 23;12:86. doi: 10.1186/1745-6215-12-86. PMID 21429214